CLINICAL TRIAL: NCT03036553
Title: The Influence of Beliefs (Fear of Movement, Pain-related Fear, Self-efficacy, and Pain Acceptance) on the Prognosis of Chronic Musculoskeletal Pain: a Prospective Cohort Study. Study Protocol
Brief Title: Influence of Beliefs on the Prognosis of Chronic Musculoskeletal Pain.
Status: Completed | Type: Observational
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Other Study IDs: UNMalaga
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2019-12

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic pain; Psychological factors; Musculoskeletal pain; Prognosis
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic musculoskeletal pain: (i) men / women over the age of 18 (ii) participants with musculoskeletal pain (pain intensity of 3 or more on a numerical scale of pain 0-10) will be included in this study, among all of the following conditions: pain around the axial skeleton (neck, lower back And / or pelvis) or peripheral joints (shoulder, elbow, wrist, knee and / or ankle). We included people with clinical diagnoses of chronic pain (shoulder pain, neck pain, whiplash disorder, temporomandibular joint disorders, pelvic pain syndrome, ankle pain and epicondylalgia), non-specific low back pain, fibromyalgia, chronic fatigue syndrome and those with a radiological diagnosis of osteoarthritis.
  (iii) duration of symptoms: more than 3 months.
  Interventions: Other: Diagnosis/Prognosis

INTERVENTIONS:
Other: Diagnosis/Prognosis — The present study will be a prospective multi-centric 12-month study that will be conducted between May 2017 and April 2019 in four primary care centers and a hospital in the province of Malaga. Several questionnaires assessing different psychological factors will be administered to these participants. The results will be evaluated at baseline (t1) and at 3-fold follow-up (after 3 (t2), 6 (t3) and 12 months (t4)).

SUMMARY:
Chronic musculoskeletal pain (CMP) is highly prevalent, disabling, and with high socio-economic costs, with many negative effects on quality of life. CMP affects the ability to perform work, social, recreational and domestic tasks, changing the mood and concentration of this population. Despite the worldwide prevalence and socioeconomic burden of CMP, a clear understanding of its etiology and pathogenesis remains elusive.

Aims:

(i) to analyze the possible level of association between pain-related fear, fear of movement, self-efficacy, and pain acceptance with pain intensity and disability at the start of the study and prospectively evaluate its predictive function; (ii) to evaluate the possible mediating role of fear of movement and self-efficacy in the relationship between pain-disability in patients with CMP.

DETAILED DESCRIPTION:
The present study will be a prospective multi-centric 12-month study that will be conducted in four primary care centers and a hospital in the province of Malaga. Several questionnaires assessing different psychological factors will be administered to these participants. The results will be evaluated at baseline (t1) and at 3 follow-up (after 3 (t2), 6 (t3) and 12 months (t4)). Ethical approval will be obtained from the Costal del Sol Ethics Committee, Malaga, Spain. This study will follow the recommendations of the Declaration of Helsinki. The study will be implemented and reported in line with the SPIRIT statement.

Participants A consecutive sample of CMP participants will be recruited. The general practitioners will carry out the recruitment. Next, the physiotherapists attending the research project, which will be previously instructed by the research team, will evaluate the participants for their eligibility. If participants meet the eligibility criteria, they will be invited to participate in this study, and then evaluated at baseline and 3, 6, and 12 months of follow-up. The inclusion criteria are: (i) men / women over the age of 18; (ii) participants with musculoskeletal pain (pain intensity of 3 or more on a numerical scale of pain 0-10) will be included in this study, among all of the following conditions: pain around the axial skeleton (neck, lower back and / or pelvis) or peripheral joints (shoulder, elbow, wrist, knee and / or ankle). We included people with clinical diagnoses of chronic pain (shoulder pain, neck pain, whiplash disorder, temporomandibular joint disorders, pelvic pain syndrome, ankle pain and epicondylalgia), non-specific low back pain, fibromyalgia, chronic fatigue syndrome and those with a radiological diagnosis of osteoarthritis. (iii) duration of symptoms: more than 3 months. Exclusion criteria are as follows: (i) musculoskeletal pain due to traumatic or systemic inflammatory autoimmune diseases such as rheumatoid arthritis, ankylosing spondylitis, spondylolisthesis or other defined rheumatological conditions; (ii) musculoskeletal pain associated with neurological dysfunction (ie, multiple sclerosis or stroke), osteoporosis, hemophilia and / or cancer; (iii) participants with post-fracture musculoskeletal pain; (iv) inability to provide informed consent and / or complete written questionnaires.

Recruitment The age and sex of those participants who refuse to participate in the project will be noted anonymously, with the objective of evaluating the external validity of the sample recruited from participants.

Eligible participants who are interested in the study will be asked to provide written informed consent to participate. Participants will complete several questionnaires at baseline, 3, 6, and 12 months after study initiation.

Participant data files will be stored in numerical order and in a safe and accessible place.

ELIGIBILITY:
Inclusion Criteria:

(i) men / women over 18 years of age; (ii) participants with musculoskeletal pain (pain intensity of 3 or more on a numerical scale of pain 0-10) will be included in this study, among all of the following conditions: pain around the axial skeleton (neck, lower back And / or pelvis) or peripheral joints (shoulder, elbow, wrist, knee and / or ankle). We included people with clinical diagnoses of chronic pain (shoulder pain, neck pain, whiplash disorder, temporomandibular joint disorders, pelvic pain syndrome, ankle pain and epicondylalgia), non-specific low back pain, fibromyalgia, Chronic fatigue syndrome and those with a radiological diagnosis of osteoarthritis. (iii) duration of symptoms: more than 3 months.

Exclusion Criteria:

(i) musculoskeletal pain due to traumatic or systemic inflammatory autoimmune diseases, such as rheumatoid arthritis, ankylosing spondylitis, spondylolisthesis or other defined rheumatological conditions; (ii) musculoskeletal pain associated with neurological dysfunction (ie, multiple sclerosis or stroke), osteoporosis, hemophilia and / or cancer; (iii) participants with post-fracture musculoskeletal pain; (iv) inability to provide informed consent and / or complete written questionnaires.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects between 18-70 years with chronic musculoskeletal pain
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline the numerical pain rating scale (NRS) at 3,6,12 months | Pain will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Pain: The Numerical Rating Scale (NRS) will assess the pain intensity of each patient at baseline and prospectively. NRS scores range from 0 to 10, with 0 without pain and 10 with the worst pain imaginable. It has been shown that the NRS has a good test-retest reliability of the same day.

SECONDARY OUTCOMES:
Change from baseline the pain disability index (PDI) at 3,6,12 months | Disability will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Disability: The Pain Disability Index (PDI) is a 7-question questionnaire that investigates the magnitude of disability due to pain in different situations such as work, leisure time, activities of daily living, and sports

OTHER OUTCOMES:
Change from baseline the tampa scale for kinsiophobia (TSK-11) at 3,6,12 months | Fear of movement will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Fear of movement: The short version of the Tampa Scale for Kinesiophobia (TSK-11) will be used to assess fear of movement
Change from baseline the fear pain questionnaire (FPQ-III) at 3,6,12 months | Pain-related fear will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Pain-related fear: The short version (9-items) of the Fear of Pain Questionnaire (FPQ-III) will be used to assess the fear of pain in this population
Change from baseline the chronic pain acceptance questionnaire (CPAQ) at 3,6,12 months | Pain acceptance will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Pain acceptance: The Chronic Pain Acceptance Questionnaire (CPAQ) will measure pain acceptance through 20 items
Change from baseline the pain self-efficacy questionnaire (PSEQ) at 3,6,12 months | Self-efficacy will be evaluated at baseline and 3 follow-ups (3,6,12 months).
  Self-efficacy: The Pain Self-Efficacy Questionnaire (PSEQ) contains 10 questions that will measure the patient's confidence in performing certain activities despite pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga
Locations (1):
- Hospital Center, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No